CLINICAL TRIAL: NCT02739945
Title: Sonographic Follow-up of Patients With Cubital Tunnel Syndrome (CTS) Undergoing Open Neurolysis in Situ or Endoscopic Release: A Prospective Study
Brief Title: Sonographic Examination Cubital Tunnel Release
Acronym: SPECTRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Marco Guidi, Dr., MD, Ente Ospedaliero Cantonale, Bellinzona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EnteOC
Record Dates: First submitted 2016-04-10; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Ulnar Nerve Compression, Cubital Tunnel
Keywords: Ulnar Nerve Compression, Cubital Tunnel
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open cubital tunnel release (Other): In situ decompression (MacKinnon and Novak 2005) is made through a 6-10 cm longitudinal incision along the course of the ulnar nerve midway between the medial epicondyle and the olecranon.
  Interventions: Procedure: Cubital tunnel release
- Endoscopic cubital tunnel release (Other): Endoscopic release follows Hoffmann's technique (Hoffmann 2006) that demonstrated the safety and efficacy of this technique in a cadaveric model and in a clinical study.
  Interventions: Procedure: Cubital tunnel release

INTERVENTIONS:
Procedure: Cubital tunnel release — The ulnar nerve is decompressed proximally at the intramuscular septum, decompressed more distally through the cubital tunnel and then exposed between the two heads of the flexor carpi ulnaris muscle. Care is taken to ensure that any point that might compress the ulnar nerve either proximally or distally is evaluated.

SUMMARY:
The investigators want to compare changes in cross-sectional area (CSA) of the ulnar nerve at the elbow after open release or endoscopic release.

DETAILED DESCRIPTION:
The investigators want to compare changes in CSA of the ulnar nerve at the elbow hypothesizing that US examination is a useful tool to detect unsuccessful release and defining which technique shows the best outcome in the first year postoperatively.

The measurement of cross-sectional area (CSA) as a diagnostic tool to detect entrapments syndrome in upper limbs has already been described. US typically demonstrates an abrupt narrowing and displacement of the nerve within the tunnel, possibly in association with a thickened retinaculum or a space-occupying lesions. Previous studies prospectively compared sonographic outcomes after decompression of the median nerve at the wrist.

ELIGIBILITY:
Inclusion Criteria:

* history of paresthesia or numbness in the ulnar nerve distribution;
* weakness or wasting of the small muscles of the hand;
* a positive elbow flexion provocation test;
* slowed motor conduction velocity in the ulnar nerve below 50 m/sec.

Exclusion Criteria:

* Patients with normal nerve conduction studies;
* prior surgery for Cubital Tunnel Syndrome;
* prior traumatic lesions of the elbow;
* coexistent neurological diseases;
* bone anormalities (cubitus valgus, deformities from previous elbow fractures, osteoarthritis with medial osteophytes ands loose bodies, heterotopic ossifications);
* subluxating ulnar nerve;
* space-occupying soft-tissue lesions.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Society Function Score | 12 months postoperatively.
  Patients undergoing surgical decompression indicate their postoperative clinical outcome with this scale

SECONDARY OUTCOMES:
Jamar dynamometer (grip strength) | 12 months postoperatively.
  Quantitative measurement of grip strength were assessed with a Jamar dynamometer. The Jamar Dynamometer is an instrument for measuring the maximum isometric strength of the hand and forearm muscles. The Jamar dynamometer was introduced in 1954 (Bechtol,1954). It consists of a sealed hydraulic system with adjustable hand spacings that measures handgrip force
Static-2 point discrimination test | 12 months postoperatively.
  Two-point discrimination is the ability to discern that two nearby objects touching the skin are truly two distinct points.
  Two-point discrimination has long been used as an assessment tool for tactile gnosis, and to assess recovery after a peripheral nerve surgery.
4-point Likert-type scale | 12 months postoperatively.
  Patients undergoing surgical decompression indicate their postoperative clinical outcome on a questionnaire using 4-point Likert-type scale (1= large improvement, 2 = moderate improvement, 3= no improvement, 4= worse than preoperatively)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Lucchina, MD, Study Director — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Dr.Lucchina Stefano, Locarno, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puig S, Turkof E, Sedivy R, Ciovica R, Lang S, Kainberger FM. Sonographic diagnosis of recurrent ulnar nerve compression by ganglion cysts. J Ultrasound Med. 1999 Jun;18(6):433-6. doi: 10.7863/jum.1999.18.6.433. No abstract available. PMID 10361850
- [Background] Martinoli C, Bianchi S, Derchi LE. Ultrasonography of peripheral nerves. Semin Ultrasound CT MR. 2000 Jun;21(3):205-13. doi: 10.1016/s0887-2171(00)90043-x. PMID 10994689
- [Background] Okamoto M, Abe M, Shirai H, Ueda N. Diagnostic ultrasonography of the ulnar nerve in cubital tunnel syndrome. J Hand Surg Br. 2000 Oct;25(5):499-502. doi: 10.1054/jhsb.1999.0350. PMID 10991822
- [Background] Watts AC, Bain GI. Patient-rated outcome of ulnar nerve decompression: a comparison of endoscopic and open in situ decompression. J Hand Surg Am. 2009 Oct;34(8):1492-8. doi: 10.1016/j.jhsa.2009.05.014. Epub 2009 Aug 20. PMID 19695795
- [Background] Hoffmann R, Siemionow M. The endoscopic management of cubital tunnel syndrome. J Hand Surg Br. 2006 Feb;31(1):23-9. doi: 10.1016/j.jhsb.2005.08.008. Epub 2005 Oct 12. PMID 16225971
- [Background] King GJ, Richards RR, Zuckerman JD, Blasier R, Dillman C, Friedman RJ, Gartsman GM, Iannotti JP, Murnahan JP, Mow VC, Woo SL. A standardized method for assessment of elbow function. Research Committee, American Shoulder and Elbow Surgeons. J Shoulder Elbow Surg. 1999 Jul-Aug;8(4):351-4. doi: 10.1016/s1058-2746(99)90159-3. PMID 10472009
- [Result] Chiou HJ, Chou YH, Cheng SP, Hsu CC, Chan RC, Tiu CM, Teng MM, Chang CY. Cubital tunnel syndrome: diagnosis by high-resolution ultrasonography. J Ultrasound Med. 1998 Oct;17(10):643-8. doi: 10.7863/jum.1998.17.10.643. PMID 9771609